CLINICAL TRIAL: NCT00369135
Title: Cross-Disciplinary Workplace Intervention Strategy for Chronic Musculoskeletal Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Universitaire Romand de Sante au Travail (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFP-111-111
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Back Pain; Neck Pain; Musculoskeletal Abnormalities
Keywords: work; Musculoskeletal Disorders
MeSH Terms: conditions — Back Pain; Neck Pain; Musculoskeletal Abnormalities; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: combined intervention

SUMMARY:
Sickness absenteeism caused by MSDs is a persistent and expensive health challenge in all industrial countries including Switzerland. Despite much progress as to the cause and prevention of MSDs, they continue to be some of the most prevalent and challenging health problems with respect to the work-place and to socio-economic burden.

To improve the situation, several recent reviews recommended interventions based on the bio-psycho-social model. Work-hardening and industrial rehabilitation programs focused more on the in balance between physical and mental demands of work on one side and capacities of the individual on the other side. Therefore we propose to merge the two models into one. The result is an interdisciplinary intervention strategy witch includes work hardening, medical trainings, a cognitive behavioural approach and work place intervention.

ELIGIBILITY:
Inclusion Criteria:

* Employees on sick leave because of non-specific back and/or neck/shoulder pain
* actual unable to work and continuous or cumulative (totalized) work incapa- city in the past 6 monts
* ≥ 20 working days 100% absence from work or
* ≥ 40 working days 80 to 99% absence from work or
* ≥ 60 working days 50 to 79% absence from work and
* not older than 58 level of employment ≥ 50%
* no longer than 6 monts absencer from work (100% unable to work)

Exclusion Criteria:

* Specific diagnosis such as infection, neoplasm, metastasis osteoporosis, rheumatoid arthritis, fracture and inflammatory process or other conditions for which valid diagnoses had been demonstrated either in the anamnesis, records or the clinical examination
* Postoperative health condition with prohibited physical load
* Major co-morbidity which may determine return to work in a clearly stronger way then the MSD itself such as a major depression, psychosis, heavy drug or alcohol disease or instable cardiac or pulmonary disease
* Predominant specific shoulder pathology in "neck-shoulder pain"

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-03; Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Sick-day saving, work capacity, economic variables | one year

SECONDARY OUTCOMES:
Functional performance, pain, general health, variables related to coping, believes, anxiety, depression | one year

CONTACTS AND LOCATIONS:
Overall Officials: Danuser Brigitta, Prof, Study Director — Institut Universitaire Romand de Sante au Travail
Locations (1):
- Institut universitaire romand de Santè au Travail, Lausanne, Switzerland

REFERENCES:
- See also: Click here for more information about this study: Cross-Disciplinary Workplace Intervention Strategy for Chronic Musculoskeletal Disorders — http://www.premus2004.ethz.ch/ZH_LAU/index.htm